CLINICAL TRIAL: NCT01138631
Title: Selection of Embryos for IVF Treatment by Time-lapse
Brief Title: Selection of Embryos by Time-lapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Professor Jakob Ingerslev, Fertility Clinic, Aarhus University Hospital, Skejby
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 25940; 25940 (Registry Identifier: Regional Ethics Comittee)
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2011-05

CONDITIONS: Infertility
Keywords: IVF, Infertility, embryo selection, embryoscope, time-lapse
MeSH Terms: conditions — Infertility | interventions — Fetoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embryoscope (Active Comparator)
  Interventions: Device: Embryoscope
- Conventional incubator (No Intervention)

INTERVENTIONS:
Device: Embryoscope — The embryoscope is an incubator with in-built photographic equipment
  Arms: Embryoscope

SUMMARY:
In order to improve success rate by assisted reproductive techniques new techniques are being developed for selection of the embryo with best chance of implantation, establishement of pregnancy and subsequent delivery.The present study is based upon the hypothesis that time-lapse (frequent imaging) may give information about important steps in embryonic development, which could help to optimize selection of embryo(s) for treatment in IVF. The present study evaluates the outcome of conventional embryo culture with culture in a specially developed incubator equipped with a time-lapse system (Embryoscope).

Embryos from 50 IVF cycles (400 embryos) will be randomised to either conventional incubation or to culture in the Embryoscope. Embryos will be cultured for five days to the blastocyst stage. The primary endpoint is fraction of embryos developed to the four cell stage.

DETAILED DESCRIPTION:
In vitro fertilization for infertility has a success rate on average in Europe of 25% in terms of baby take-home rate per cycle. One way to improve this rather low succes rate is to develop new measures for selection of the best embryo among peers as presently evaluated by embryo morphology. One of these promising methods is contineous imaging of embryo development by time-lapse. A new and unique equipment for this purpose - an Embryoscope - har been developed by Unisense Fertilitech. The present study evaluates embryo 4-cell rate during cultivation to blastocyst stage in a conventional incubator with 4-cell rate in the Embryoscope to ensure non-inferiority of the latter.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing 2.nd or 3.rd IVF cycle with expected retrieval of 8 oocytes or more. Age < 38 years

Exclusion Criteria:

* Endometriosis

Max Age: 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
4-cell rate | 2 days after oocyte pick-up

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Ingerslev, DMSc, Principal Investigator — University of Aarhus
Locations (1):
- Fertility Clinic, Aarhus University Hospital, Skejby, Aarhus, Aarhus, Denmark